CLINICAL TRIAL: NCT06793501
Title: A Reablement Intervention in Residential Aged Care (Re-RAC): Study Protocol for a Multi-center, Pragmatic Randomized Controlled, Open-label Trial
Brief Title: Reablement in Residential Aged Care - a Randomized Controlled Trail
Acronym: Re-RAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Kajsa Lidström Holmqvist, Associate professor, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 282513
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Older People
MeSH Terms: interventions — Control Groups; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reablement intervention (Experimental): Participants recieve reablement intervention
  Interventions: Other: Reablement intervention
- Control group (Active Comparator): Participants recieve treatment as usual which is conventional care
  Interventions: Other: Control group

INTERVENTIONS:
Other: Reablement intervention — Reablement's implementation in this study is characterized by a comprehensive assessment of the older person's everyday activities, both current and past. This is done through a person-centered interview using the Canadian Occupational Performance Measure (COPM). The COPM is based on the assumptions described in the theoretical framework of CMOP-E. Based on the assessment, the older adult selects a personal activity goal, which consists of an activity they consider meaningful and wish to improve. In collaboration with the older adult and staff, a goal-oriented support plan, also referred to as a training program, is developed to achieve the goal. Nursing assistant staff support the older persons in performing defined training activities and receive supervision from rehabilitation staff. The support plan and progress toward the activity goal are evaluated through regular reassessments during a fixed intervention period of eight weeks.
  Other Names: Re-RAC
  Arms: Reablement intervention
Other: Control group — TAU includes a general approach where all activities that the older adult engages in during everyday life are considered rehabilitative. The staff are encouraged to motivate the older adult to do as much as possible independently, in order to prevent loss of function and maintain the ability to perform activities. The approach does not involve any direction toward specific activities where there is a rehabilitative need. It does not include any formulated goals or follow-up. Additionally, there is no specific education offered to the nursing assistants on how to encourage the older adult or how to follow-up up on the extent to which the approach is applied.
  Other Names: Treatment as usual
  Arms: Control group

SUMMARY:
Background: The global increase in older adults presents challenges for maintaining health and autonomy in residential aged care (RAC) facilities, where passivity has been shown to often diminish quality of life. However, the reablement approach, which enhances independence through personalized, multidisciplinary strategies, shows promise for addressing these issues and requires further evaluation, particularly in Swedish contexts.

The research project Reablement in RAC (Re-RAC) aims to evaluate the impact of the Re-RAC intervention on activity performance and satisfaction, participation, quality of life and well-being, and health economic outcomes for older adults in RAC facilities, while also describe participant and staff experiences.

Methods: This study is a multi-center prospective pragmatic randomized controlled trial with two parallel groups that will evaluate the Re-RAC intervention compared to treatment as usual, using quantitative, qualitative and health economic methods.

The Re-RAC intervention begins with an interview according to Canadian Occupational Performance Measure (COPM) to identify a meaningful goal, followed by a personalized support plan with training activities, supported by nursing staff. The intervention lasts 8 weeks, with adjustments made based on progress, and ends with a COPM reassessment of the participant's performance and satisfaction. Eighty-six participants will be included, assessed for performance (COPM-performance), satisfaction (COPM-satisfaction), health-related quality of life (EQ-5D-5L), psychological well-being (WHO-5), and physical activity levels (measured by an accelerometer), before and after the intervention. Pain will also be assessed for potential associations with other outcomes. Participants' and staff's experiences will be described through interviews, and cost-effectiveness will be evaluated by calculating the cost per quality adjusted life-years gained.

Discussion: The Re-RAC project evaluates the impact of a reablement intervention on activity performance, satisfaction, quality of life, well-being, and health outcomes for older adults in RAC facilities through a pragmatic randomized controlled trial, with assessments before and after the 8-week intervention. The study also explores participant and staff experiences and evaluates cost-effectiveness. The results of this study will offer valuable insights to inform the future implementation and assessment of reablement interventions in RAC settings.

ELIGIBILITY:
Inclusion Criteria: Older adults aged 65 years and above, residing in a somatic ward at one of the RAC facilities where the study will be conducted, and meeting the inclusion criteria, are eligible to participate in the study. The inclusion criteria require that the older adult must be able to engage in conversations in Swedish and be able to participate in both the assessments and the intervention.

Exclusion Criteria: Persons having severe cognitive impairment (≤17) according to Mini Mental State Examination-Swedish version (MMSE-SR; screening for cognitive function) or being very severely frail or terminally ill according to Clinical Frailty Scale (≥8) (CFS-9) will be excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in occupational performance related to the prioritized activity, measured with the COPM-P | From enrollment to the end of treament after 8 weeks
  The COPM is an interview-administered instrument used to assess occupational performance (COPM-P) and satisfaction with performance (COPM-S) for up to five self-determined activity issues in the areas of self-care, productivity, and leisure. Participants will rate their performance and satisfaction with their highest-priority activity on a scale of 1-10, where 1 = unable to perform at all/not satisfied at all, and 10 = able to perform extremely well/extremely satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Care Research Center, Örebro, Örebro County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Philipson A, Lindvall MA, Pettersson C, Stralman L, Holmqvist KL. Reablement in Residential Aged Care (Re-RAC): study protocol for a multi-center pragmatic randomized controlled open-label trial. Trials. 2025 Aug 18;26(1):294. doi: 10.1186/s13063-025-08999-0. PMID 40826363